CLINICAL TRIAL: NCT02916121
Title: Relationships of One-carbon Cycle Pathway With Psychopathology and Metabolic Abnormalities in Patients With Schizophrenia and Potential Intervention Strategy With Folic Acid and Vitamin B12
Brief Title: Potential Intervention Strategy With Folic Acid and Vitamin B12 in Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201408009
Record Dates: First submitted 2016-08-29; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Folic Acid; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- folic acid 5 mg/cap (Experimental): folic acid 5 mg/d and vitamin B12 500 ug/d
  Interventions: Dietary Supplement: folic acid 5 mg/cap
- placebo (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: folic acid 5 mg/cap — the intervention includes folic acid 5 mg/d and vitamin B12 500 ug/d
  Other Names: vitamine B12 500 ug/cap
  Arms: folic acid 5 mg/cap
Other: Placebo — placebo
  Arms: placebo

SUMMARY:
The investigators study aims are:

1. To investigate folate, vitamin B12, and homocysteine levels in patients with schizophrenia.
2. To evaluate the relationships among folate, vitamin B12, and homocysteine levels, genetic variants of one-carbon cycle pathway, psychopathology, including positive symptoms, negative symptoms, and cognition, and metabolic abnormalities in patients with schizophrenia.
3. For patients with low folate levels, the investigators would like to conduct a 24-week double-blinded, placebo-controlled of folic acid (5 mg/d) and vitamin B12 (500 ug/d) supplementation study to know whether combination of folic acid and vitamin B12 can improve patients' psychopathology or metabolic profiles, and the effects of genetic variants in one-carbon cycle pathway on treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-65 year-old.
2. Fulfill DSM-IV-TR diagnosis of schizophrenia.
3. Be treated with an antipsychotic agent for at least 6 months or at a stable dose for at least 3 months.
4. Patients with folate deficiency or insufficiency, and PANSS score at least 60 or more in the first phase screening.

Folate deficiency and insufficiency (low folate level) are defined as serum folate < 6.8 nmol/L (3 ng/mL) and <= 13.5 nmol/L (6 ng/mL), respectively.

Exclusion Criteria:

1. Medically unstable.
2. Currently taking vitamin supplementation.
3. Pregnancy or lactation.
4. Test positive of urine drug screen
5. Megaloblastic anemia due to folate deficiency;
6. Patients with parkinsonism (score of > 12 on the Simpson-Angus Scale);
7. History of alcohol or other substances use disorder in past 3 months;
8. History of significant neurological illness;
9. Creatine>1.4 ng/dl.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 24 weeks
  We used PANSS to evaluate patients' psychopathology at baseline, week-2, 4, 8, 12, 16, 20, and 24.

SECONDARY OUTCOMES:
CogStat neuropsychological test, including speed of processing, attention, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition | 24 weeks
  CogStat will be used to test patients' cognitive function, including speed of processing, attention, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition, at baseline and week-24.
blood pressure, mmHg | 24 weeks
  Blood pressure will be checked at week 4, 12, and 24.
waist circumference, cm | 24 weeks
  Waist circumference will be checked at week 4, 12, and 24.
triglyceride, mg/dL | 24 weeks
  Triglyceride will be checked at week 4, 12, and 24.
high density lipoprotein cholesterol (HDL-C), mg/dL | 24 weeks
  HDL-C will be checked at week 4, 12, and 24.
fasting blood sugar level, mg/dL | 24 weeks
  fasting blood sugar level will be checked at week 4, 12, and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Hsin Chen, MD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided